CLINICAL TRIAL: NCT03023839
Title: Incidence and Risk Factors for Delirium in Severely Injured Patients
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyung, associate professor, Asan Medical Center
Other Study IDs: 2014-0344
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Delirium; Trauma; Intensive Care Unit Syndrome
Keywords: Delirium; Trauma; Injury; restraints
MeSH Terms: conditions — Delirium; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe trauma patients: Severe Trauma patients (ISS >15) admitted to Intensive Care Unit (ICU)

SUMMARY:
Delirium is very common in intensive care unit (ICU) patients and leads to poor outcomes. There is little information on delirium in injured patients however. This study determined the incidence and risk factors for delirium in severely injured patients.

DETAILED DESCRIPTION:
This study was a prospective cohort study that reviewed the medical records of 179 trauma patients who were admitted to Asan Medical Center from January 01, 2013 to December 31, 2014. The investigators included all patients who had an Injury Severity Score (ISS) of more than 15 and excluded patients younger than 15 years old. This study was approved by the Asan Medical Center Institutional Review Board (2014-0344).

Patient delirium was checked using the Confusion Assessment Method in Intensive Care Unit (CAM-ICU) three times every day. The CAM-ICU includes four features that assess acute changes in or the fluctuating course of mental status, inattention, altered level of consciousness, and disorganized thinking. If a patient has a Richmond Agitation Sedation Scale (RASS) score of -3 or more with acute changes in mental status, inattention, and disorganized thinking or altered level of consciousness, a diagnosis of delirium can be made. The investigators considered patients to be delirious when CAM-ICU was positive for more than 24 h.

The investigators reviewed clinical information for the study patients including age, sex, and underlying disease. Trauma factors reviewed were cause of trauma, ISS, Glasgow Coma Scale (GCS) score, shock, initial lactate level, massive transfusion within 24 h, cardiopulmonary resuscitation rescue, and time taken to the hospital after trauma. Factors related to treatment included use of restraints, mechanical ventilation, and surgery. Clinical outcomes included mortality, ICU stay, mechanical ventilation duration, and hospital stay.

Statistical analysis were done using both univariate (chi-square test and t-test) and multivariate (logistic regression) procedures. Results are reported as mean ± standard deviation. Significance set at a P value of less than .05. For the multivariable logistic regression, the primary outcome variable of interest was the development of delirium after trauma that was classified as either present or absent. Variables were entered for analysis based on the strength of their univariate association with the presence/absence of delirium.

ELIGIBILITY:
Inclusion Criteria:

* trauma patients with Injury Severity Score (ISS) more than 15

Exclusion Criteria:

* age under 15

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe Trauma patients admiited to Intensive Care Unit (ICU) of Asan Medical Center from 01 Jan 2013 to 31 Dec 2014
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium in trauma patients | within the 6 months after ICU admission
risk factors of delirium in trauma patients | within the 6 months after ICU admission

SECONDARY OUTCOMES:
hospital stay of delirium in trauma patients | within the 6 months after ICU admission
ICU stay of delirium in trauma patients | within the 6 months after ICU admission
mechanical ventilation days of delirium in trauma patients | within the 6 months after ICU admission
mortality of delirium in trauma patients | within the 6 months after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Suk-kyung Hong, Ph.D, Principal Investigator — University of Ulsan College of Medicine. Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reade MC, Finfer S. Sedation and delirium in the intensive care unit. N Engl J Med. 2014 Jan 30;370(5):444-54. doi: 10.1056/NEJMra1208705. No abstract available. PMID 24476433
- [Background] Angles EM, Robinson TN, Biffl WL, Johnson J, Moss M, Tran ZV, Moore EE. Risk factors for delirium after major trauma. Am J Surg. 2008 Dec;196(6):864-9; discussion 869-70. doi: 10.1016/j.amjsurg.2008.07.037. PMID 19095101
- [Background] Thomason JW, Shintani A, Peterson JF, Pun BT, Jackson JC, Ely EW. Intensive care unit delirium is an independent predictor of longer hospital stay: a prospective analysis of 261 non-ventilated patients. Crit Care. 2005 Aug;9(4):R375-81. doi: 10.1186/cc3729. Epub 2005 Jun 1. PMID 16137350
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Pandharipande P, Cotton BA, Shintani A, Thompson J, Pun BT, Morris JA Jr, Dittus R, Ely EW. Prevalence and risk factors for development of delirium in surgical and trauma intensive care unit patients. J Trauma. 2008 Jul;65(1):34-41. doi: 10.1097/TA.0b013e31814b2c4d. PMID 18580517
- [Background] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Background] Gani H, Domi R, Kodra N, Prifti P, Naco M, Beqiri V, Torba D, Tare R. The incidence of postoperative delirium in elderly patients after urologic surgery. Med Arch. 2013;67(1):45-7. doi: 10.5455/medarh.2013.67.45-47. PMID 23678839
- [Background] Cavallazzi R, Saad M, Marik PE. Delirium in the ICU: an overview. Ann Intensive Care. 2012 Dec 27;2(1):49. doi: 10.1186/2110-5820-2-49. PMID 23270646
- [Background] Mistraletti G, Carloni E, Cigada M, Zambrelli E, Taverna M, Sabbatini G, Umbrello M, Elia G, Destrebecq AL, Iapichino G. Sleep and delirium in the intensive care unit. Minerva Anestesiol. 2008 Jun;74(6):329-33. PMID 18500209
- [Background] Brummel NE, Girard TD. Preventing delirium in the intensive care unit. Crit Care Clin. 2013 Jan;29(1):51-65. doi: 10.1016/j.ccc.2012.10.007. PMID 23182527